CLINICAL TRIAL: NCT01849185
Title: Probiotic BIO-25 as a Supplement to Statins for the Treatment of Hypercholesterolemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mmc120213ctil
Record Dates: First submitted 2013-05-05; First posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIO 25 (food supplements)twice a day for 8 weeks (Active Comparator): BIO 25 - Innovative Formula contains 11 different strains of probiotic bacteria patents and more than 25 billion active bacteria in each capsule.
  Interventions: Other: Food supplement
- Placebo twice a day for 8 weeks (Placebo Comparator): Placebo twice a day for 8 weeks
  Interventions: Other: Food supplement

INTERVENTIONS:
Other: Food supplement
  Other Names: BIO-25

SUMMARY:
The primary objective is to examine whether probiotics given to hypercholesterolemic patients treated with statins, would further decrease LDL-Cholesterol levels.

The secondary objective is to examine whether adding of probiotics to statins would decrease fasting glucose levels and glycolysated hemoglobin

ELIGIBILITY:
Inclusion Criteria:

1) Patients on maximal tolerated dose of conventional statins treated for at least eight weeks on simvastatin 40, pravastatin 40, atorvastatin 40-80 or rosuvastatin 20-40 mg, who failed to achieve target values of LDL-cholesterol according to the European Socety Cardiology guidelines 2012.

Exclusion Criteria:

1. Patients on chronic antibiotic treatment
2. Patients with immune disorders
3. Patients who are not receiving maximal dose of statin therapy or receive combination of statins for dyslipidemia.
4. Patients who experienced myocardial infarction within less than two months.
5. Patients who consume probiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-01 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
LDL-Cholesterol levels. | 8 weeks
  The primary objective is to examine whether probiotics given to hypercholesterolemic patients treated with statins, would further decrease LDL-Cholesterol levels.

SECONDARY OUTCOMES:
Hemoglobin A1C | 8 weeks
  The secondary objective is to examine whether adding of probiotics to statins would decrease fasting glucose levels and glycosylated hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Berlin, MD, Principal Investigator — Division of Cardiology Meir MC
Locations (1):
- Division of Cardiology Meir MC, Kfar Saba, Israel